CLINICAL TRIAL: NCT06494319
Title: Development Of a Virtual Stress Inoculation Training (SIT) Platform and Mobile Health App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sarah Jackson, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0547
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: PTSD; Trauma and Stressor Related Disorders; Traumatic Brain Injury
Keywords: veteran; Post Traumatic Stress Disorder (PTSD); Traumatic Brain Injury; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The first 10 participants will do the treatment via the canvas classroom virtually and participate in user experience interviews to improve the quality of the treatment and improve the user experience.Next, the second group of 10 participants will do the treatment with the canvas classroom aided by a mobile health application.These participants will also participate in user experience interviews to improve the quality of the treatment and improve the user experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIT NAVIGATOR plus Stress NAVIGATOR group (Experimental)
  Interventions: Behavioral: Stress NAVIGATOR (Mobile Health Application); Behavioral: SIT NAVIGATOR
- SIT NAVIGATOR only group (Active Comparator)
  Interventions: Behavioral: SIT NAVIGATOR

INTERVENTIONS:
Behavioral: Stress NAVIGATOR (Mobile Health Application) — Participants will be prompted to complete their assessments each week (or upon completion of each session) via the Stress NAVIGATOR mobile health app
  Arms: SIT NAVIGATOR plus Stress NAVIGATOR group
Behavioral: SIT NAVIGATOR — Participants will complete 11 self-paced virtual SIT sessions in the SIT-NAVIGATOR classroom. Participants will be asked to complete at least one session per week, in a minimum of 12 weeks and a maximum of 14 weeks.

SUMMARY:
The purpose of this study is to demonstrate the feasibility and utility of SIT delivered asynchronously (self-paced) via fully virtual platform with and without the aid of a mobile health application and to determine initial change over baseline in terms of reduction in PTSD symptoms and improvement in resiliency in participants receiving the virtual SIT prototype, using Linear Mixed Models (LMMs),

ELIGIBILITY:
Inclusion Criteria:

* US Military Veterans / Service Members
* diagnosis of PTSD as measured by a Posttraumatic Symptom Checklist for DSM-5 (PCL-5) score of >33
* history of combat trauma and/or military service in an imminent danger pay area
* be fluent in English.
* be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
* have access to a SmartPhone or tablet to utilize the mobile health app and/OR access the virtual classroom.
* agree to undergo psychometric testing and participate in ongoing assessments throughout the study duration.
* be willing to comply with all study procedures, able to complete all assessments independently, and available for the duration of the study.

Exclusion Criteria:

* Active suicidal ideation as assessed by the Investigator at screening or as identified during the study.
* Clinically significant history of psychotic disorder, bipolar spectrum disorder, or neurodegenerative disease/dementia as assessed by the Investigator.
* Active severe substance abuse as assessed by the investigator in accordance with DSM-5 Substance Abuse Disorder criteria, an AUDIT score > 15, or partial Brief Addiction Monitor (BAM) indicating the presence of illicit substance use other than cannabis (< 3 times weekly).
* They are currently undergoing another form of treatment other than supportive therapy (> 2 times per month).
* Engaged in active trauma-focused therapy including Cognitive Processing Therapy (CPT)Prolonged Exposure (PE), or Eye Movement Desensitization and Reprocessing (EMDR).
* Any other condition/situation that the Investigator believes may interfere with participant safety, study conduct, or interpretation of study data.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduced symptoms of PTSD as assessed by the Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) | end of study (about 11-14 weeks after baseline)
  This is a 20 item questionnaire , each is scored from 0(not at all) -4( extremely)for a maximum score of 80, higher score indicating worse outcome
Increasing resilience as assessed by The Connor-Davidson Resilience Scale-10 (CD-RISC-10)4 | end of study (about 11-14 weeks after baseline)
  This is a 10 item questionnaire , each is scored from 0(not true at all) to 4(true nearly all the time) for a maximum score of 40, higher score indicating better outcome
Satisfaction with care as assessed by the Client Satisfaction Questionnaire-8-item (CSQ-8) | 4 weeks after baseline
  This is an 8 item questionnaire , each is scored on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied,poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent). for a score range of 8-32, higher score indicating better outcome
Satisfaction with care as assessed by the Client Satisfaction Questionnaire-8 item ( CSQ-8) | 8 weeks after baseline
  This is an 8 item questionnaire , each is scored on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied,poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent). for a score range of 8-32, higher score indicating better outcome
Satisfaction with care as assessed by the Client Satisfaction Questionnaire (8-item; CSQ-8) | end of study (about 11-14 weeks after baseline)
  This is an 8 item questionnaire , each is scored on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied,poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent). for a score range of 8-32, higher score indicating better outcome
Change in average heart rate as assessed by the emWave Inner Balance personal biofeedback device by HeartMath | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  Heart rate is measured in beats per minute
Change in average coherence(heart rate variability) as assessed by the emWave Inner Balance personal biofeedback device by HeartMath | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  Heart rate variability is measured via a mathematical algorithm called coherence
Change in achievement score as assessed by the emWave Inner Balance personal biofeedback device by HeartMath | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  Achievement is measured via mathematical equation that includes coherence and heart rate variability and beats per minute over time. Higher achievement is associated with higher coherence sustained over time.
Patient satisfaction as assessed by the Client Satisfaction Questionnaire (8-item; CSQ-8) | 4-6 weeks(mid treatment)
  The CSQ-8 is an 8-item measurement of global satisfaction. The range of possible scores is 8-32; higher scores indicate higher satisfaction with treatment. Items are measured on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied, poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent).
Patient satisfaction as assessed by the Client Satisfaction Questionnaire (8-item; CSQ-8) | 6-8 weeks (mid treatment)
  The CSQ-8 is an 8-item measurement of global satisfaction. The range of possible scores is 8-32; higher scores indicate higher satisfaction with treatment. Items are measured on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied, poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent).
Patient satisfaction as assessed by the Client Satisfaction Questionnaire (8-item; CSQ-8) | end of treatment (11-14 weeks)
  The CSQ-8 is an 8-item measurement of global satisfaction. The range of possible scores is 8-32; higher scores indicate higher satisfaction with treatment. Items are measured on a 4-point Likert scale where 1 indicates low satisfaction with care (e.g., quite dissatisfied, poor) and 4 indicates high satisfaction with care (e.g., very satisfied, excellent).

SECONDARY OUTCOMES:
Change in difficulty to fall sleep as assessed by the Insomnia Severity Index (ISI) | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  This is a 7 item questionnaire, with a score range from 0-28, higher score indicating more insomnia
Change in severity of depression as assessed by the Patient Health Questionnaire (PHQ-9) | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) for a maximum score of 27, higher score indicating worse outcome
Change in pain interference as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)-Pain Interference scale | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  This is a 6 item questionnaire and each is scored from 1(not at all) to 5(very much) for a maximum score of 30, higher score indicating more pain interference
Change in pain intensity as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)-Pain Intensity scale | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  This is a 3 item questionnaire and each is scored from 1(had no pain) to 5(severe pain) for a maximum score of 15, higher score indicating more pain
Change in adaptability to stress as assessed by the Situational Adaptation to Stress Scale (SASS-HSR) | Baseline , 4-6 weeks(mid treatment), end of treatment (11-14 weeks)
  This is an 18 item questionnaire and each is scored from 1( totally disagree) to 5 (agree) for a maximum score of 90, higher score indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jackson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No